CLINICAL TRIAL: NCT03065270
Title: Efficacy of Masai Barefoot Technology (MBT) for Decreasing Pain and Improvement of Lumbopelvic Pain
Brief Title: Efficacy of Unstable Shoes for Instability and Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Raquel Díaz-Meco Conde, Principal Investigador, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEM-DOL-2011-01
Record Dates: First submitted 2017-02-10; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Lumbopelvic Postpartum Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental)
  Interventions: Other: Use unstable shoes Masai Barefoot Technology (MBT)
- B group (Experimental)
  Interventions: Other: Use conventional sport shoes

INTERVENTIONS:
Other: Use unstable shoes Masai Barefoot Technology (MBT) — Use of unstable shoes during 9 weeks, at least four hours per day.
  Arms: A group
Other: Use conventional sport shoes — Use of conventional sport shoes during 9 weeks, at least four hours per day.
  Arms: B group

SUMMARY:
During pregnancy, pregnant women adopt an atypical pattern position with the intention to maintain stability and balance.These postural changes can cause instability at the level of the sacroiliac joint with painful condition during pregnancy and postpartum.

40 % of women have postpartum lumbopelvic instability. In 17 % of cases the lumbopelvic pain is perpetuated.

Another alteration influenced by the gestational status and progress of labor is urinary incontinence (UI).

The mechanism developed by Masai Barefoot Technology (MBT) provides an unstable base. Some studies reviewed, indicate that this shoe increases muscle activity, contributes to the decrease of joint overload and thereby, decreases pain.

Objective To compare the efficacy of shoes with unstable sole MBT®, over the use of conventional sports shoes, in primiparous women with lumbopelvic postpartum pain.

Material and Methods Randomized clinical trial. 24 postpartum women from the Gynecology Service of the Hospital Universitario Madrid Chiron were included in the study.

The subjects were randomly divided into experimental and control group.

ELIGIBILITY:
Inclusion Criteria:

Primparous women.

* Postpartum, between 8-12 weeks after the date of delivery.
* With lumbopelvic pain and positive diagnostic tests of sacroiliac pain
* Women with ambulation ability.

Exclusion Criteria:

* Presence of vaginal prolapses.
* Be receiving another treatment for the alteration that concerns us, pharmacological or any other type of therapy.
* Neuromuscular alterations.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pain | 9th week
  Sacroiliac pain provocation test.

SECONDARY OUTCOMES:
Pelvic Stability | 9th week
  Podiatric Stabilometry.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Diaz-Meco Conde, Doctor, Principal Investigator — Universidad Europea

IPD SHARING:
Plan to Share IPD: No